CLINICAL TRIAL: NCT06563726
Title: Partnering With Parents for Pumping Success: Feasibility of Personalized Lactation Support Utilizing Point-of-Care Human Milk Biomarkers
Brief Title: Sodium Awareness in Lactation Trial
Acronym: SALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Samantha Anthony, Health Clinician Scientist, Associate Professor, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PJM-185757
Record Dates: First submitted 2024-08-08; First posted 2024-08-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Breastfeeding; Preterm Birth; Breast Pumping; Lactation; Insufficient, Partial
MeSH Terms: conditions — Breast Feeding; Premature Birth; Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: multi-centre, non-blinded, non-randomized prospective interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: point-of-care milk sodium testing — Data-driven interventions to improve early lactation success are lacking, and parents who deliver preterm are at high risk of lactation challenges. We will be studying feasibility, acceptability, and time cost of teaching lactating parents of hospitalized preterm infants how to test their breastmilk sodium (Na) using point-of-care (POC) meters. As a secondary aim, we will assess the potential to use these POC sodium results to guide personalized lactation care in the form of altered pumping schedules in an attempt to reduce breastmilk Na. A drop in Na is a sign of secretory activation in the breast that is associated with adequate short and long-term breast milk volumes in this vulnerable population.

SUMMARY:
SALT is a multi-centre, non-blinded, non-randomized prospective interventional pilot study teaching lactating parents of hospitalized preterm infants how to test their breastmilk sodium (Na) using point-of-care (POC) meters. A drop in Na is a sign of secretory activation in the breast that is associated with adequate short and long-term breast milk volumes in this vulnerable population.

Primary Objective: Establish feasibility, acceptance, and time cost of parent-led parent milk Na testing in the first 14 days postpartum

Secondary Objective: Further investigate relationships between pumping behaviours, lactation risk factors, daily milk Na and lactation outcomes

Exploratory Objective: Explore how POC Na data may be used to modify pumping behaviour and milk volumes

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Have delivered a preterm singleton or twin infant at <35 weeks gestation admitted to a study NICU at birth or transferred into a study NICU from another NICU within the first 72 hours postpartum
3. Day 5 or less postpartum (Day 1 = day of delivery) upon enrollment (ideally day 3 or less)
4. Plans to lactate at least 2 weeks and initiate lactation with a breast pump
5. Expected infant NICU stay of 7+ (ideally 14+) days in enrollment NICU(s)

Exclusion Criteria:

1. Potential study participant's infant is critically ill and not expected to survive or has lethal diagnosis with plans by medical team/family to redirect care
2. Has delivered triplets or higher order multiples (potential confounder for lactation challenges; of note, triplets or higher are rare, on the order of a few parents annually)
3. Lactation contraindication(s) (i.e., active chemotherapy) or declines lactation initiation
4. History of breast surgery that may affect ability to lactate (i.e., breast reduction; breast augmentation that utilized nipple incisions)
5. Using or planning to use hormonal birth control in the first 14 days post-partum as may affect secretory activation/lactation
6. Unable/unwilling to be present in study NICU during any of first 5 days postpartum
7. Presumption by the medical team that infant will be in study NICU for <5 days

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Establish feasibility of parent-led longitudinal parent milk Na testing in the first 14 days postpartum: economic | First 14 days postpartum
  We will collect time cost of milk testing, including teaching parents how to test milk and daily time testing milk. This outcome will include time (in hours) spent in the first 14 days for parent and staff, with a health economist determining costs for that time
Establish feasibility of parent-led longitudinal parent milk Na testing in the first 14 days postpartum: parent acceptance via interviews | First 14 days postpartum
  We will collect qualitative data on parent acceptance and feelings about Na testing from parent interviews
Establish feasibility of parent-led longitudinal parent milk Na testing in the first 14 days postpartum: parent acceptance via surveys | First 14 days postpartum
  We will collect qualitative data on parent acceptance and feelings about Na testing from parent surveys

SECONDARY OUTCOMES:
Investigate inter-relationships between pumping frequency, parent lactation risk factors, daily milk Na levels and longer term lactation outcomes (milk provision at NICU discharge). | Enrollment to infant NICU discharge, up to 52 weeks (average NICU stay is about 10 weeks)
  We will assess interrelationships between aforementioned factors and milk provision at NICU discharge (exclusive, any, none). Note these are not necessarily correlations, but relationships and associations that we will analyze and explore in various models and combinations, so these outcome cannot be separated.
Investigate inter-relationships between pumping frequency, parent lactation risk factors, daily milk Na and short term lactation outcomes (coming to volume) | First 14 days postpartum
  We will assess interrelationships between aforementioned factors and coming to volume (pumping at least 500mL/day by postpartum day 14).Note these are not necessarily correlations, but relationships and associations that we will analyze and explore in various models and combinations, so these outcomes cannot be separated.

OTHER OUTCOMES:
Explore if POC Na data used to recommend changes in pumping behaviour is associated with actual changes in parent pumping behaviour | First 14 days postpartum
  Explore in parents whom we recommend to modify pumping frequency, rates of coming to volume by day 14 (pumping at least 500mL/day)
Explore how POC Na data used to recommend changes in pumping behaviour is associated with short-term milk volumes | First 14 days postpartum
  Determine in parents whom we recommend to modify pumping frequency based on POC Na, how often they actually followed our recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J. Anthony, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- United States (2):
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT06563726/Prot_SAP_000.pdf